CLINICAL TRIAL: NCT05314842
Title: Clinical and Radiographic Evaluation of Pulpotomy in Primary Molars Treated With Premixed Bio-ceramic MTA Versus Formocresol Among a Group of Egyptian Children: A Pilot Study.
Brief Title: Pulpotomy in Primary Molars Treated With Premixed Bio-ceramic MTA Versus Formocresol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarah Abdelbar Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Sarah Abdelbar Mahmoud, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 203
Record Dates: First submitted 2022-03-25; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Caries
MeSH Terms: interventions — formocresol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): the group that have caries in primary molars and treat them with formocresol
  Interventions: Drug: Formocresol
- experimental group (Experimental): the group that have caries in primary molars and treat them with premixed bioceramic MTA
  Interventions: Drug: Premixed bioceramic MTA

INTERVENTIONS:
Drug: Formocresol — dressing agents in pulpotomized primary molas using formocresol in cariously exposed vital primary molars
  Arms: control group
Drug: Premixed bioceramic MTA — dressing agents in pulpotomized primary molas using premixed bioceramic MTA in cariously exposed vital primary molars
  Other Names: Neoputty
  Arms: experimental group

SUMMARY:
examine the results of pulpotomy in primary molars using premixed bioceramic MTA versus Formocresol. Clinical and radiographic success rates were used as outcomes.

DETAILED DESCRIPTION:
Primary outcome:

Soft-tissue pathology

* Post-treatment swelling will be assessed through visual examination by the operator, either intraorally or extra orally.
* Sinus tract or fistula will be assessed through visual examination by the operator

Secondary outcomes:

1. Pain to the percussion will be assessed by gentle tapping on the tooth with the end of a dental mirror
2. mobility will be assessed through the back of two mirrors
3. radiographic assessments:- for any radiolucency and pathologic root resorption (periapical or bifurcation) will be examined (present or not).

clinical assessment on every recall visit during the 3-, 6-, and 12-month follow-up period.

• These radiographic assessments will be performed as baseline data at the first visit following the operating procedure, as well as at 3, 6, and 12 months after the baseline.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit and cooperative children.
* Pediatric patients aged 4-6 years.
* A deep carious lesion in vital primary molars.
* Absence of clinical signs and symptoms of pulpal exposure.
* Absence of radiographic signs and symptoms of people degeneration.
* Positive parental informed consent.

Exclusion Criteria:

Uncooperative children.

* Medically compromised children.
* Presence of clinical signs and symptoms of pulpal exposure.
* Presence of radiographic signs and symptoms of pulp degeneration.
* Physiologic root resorption more than one-third.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Soft-tissue pathology | at 0 day
  * Post-treatment swelling will be assessed through visual examination by the operator, either intraorally or extra orally.
  * Sinus tract or fistula will be assessed through visual examination by the operator.
  Binary (present or absent)
Soft-tissue pathology | at 3 month
  * Post-treatment swelling will be assessed through visual examination by the operator, either intraorally or extra orally.
  * Sinus tract or fistula will be assessed through visual examination by the operator.
  Binary (present or absent)
Soft-tissue pathology | at 6 month
  * Post-treatment swelling will be assessed through visual examination by the operator, either intraorally or extra orally.
  * Sinus tract or fistula will be assessed through visual examination by the operator.
  Binary (present or absent)
Soft-tissue pathology | at 1 year
  Post-treatment swelling will be assessed through visual examination by the operator, either intraorally or extra orally.
  -Sinus tract or fistula will be assessed through visual examination by the operator.
  Binary (present or absent)

SECONDARY OUTCOMES:
• Pain to the percussion | at 0 day
  will be assessed by gentle tapping on the tooth with the end of a dental mirror.
  Binary (present or absent)
• Pain to the percussion | at 3 month
  will be assessed by gentle tapping on the tooth with the end of a dental mirror.
  Binary (present or absent)
• Pain to the percussion | at 6 month
  will be assessed by gentle tapping on the tooth with the end of a dental mirror.
  Binary (present or absent)
• Pain to the percussion | at 1 year
  will be assessed by gentle tapping on the tooth with the end of a dental mirror.
  Binary (present or absent)
mobility | at 0 day
  • Mobility is scored on a scale of 1-3 as follows:
  1. the movement that is greater than normal (physiological) movement.
  2. a maximum of 1 mm in the buccolingual direction.
  3. depreciable buccolingual movement of more than 1 mm. Miller's Grades
mobility | at 3 month
  • Mobility is scored on a scale of 1-3 as follows:
  1. the movement that is greater than normal (physiological) movement.
  2. a maximum of 1 mm in the buccolingual direction.
  3. depreciable buccolingual movement of more than 1 mm. Miller's Grades
mobility | at 6 month
  • Mobility is scored on a scale of 1-3 as follows:
  1. the movement that is greater than normal (physiological) movement.
  2. a maximum of 1 mm in the buccolingual direction.
  3. depreciable buccolingual movement of more than 1 mm. Miller's Grades
mobility | at 1 year
  • Mobility is scored on a scale of 1-3 as follows:
  1. the movement that is greater than normal (physiological) movement.
  2. a maximum of 1 mm in the buccolingual direction.
  3. depreciable buccolingual movement of more than 1 mm. Miller's Grades
radiographic indications of radiolucency and pathologic root resorption (periapical or bifurcation) will be examined (present or not). | at 0 day
  Binary (present or absent)
radiographic indications of radiolucency and pathologic root resorption (periapical or bifurcation) will be examined (present or not). | at 3 month
  Binary (present or absent)
radiographic indications of radiolucency and pathologic root resorption (periapical or bifurcation) will be examined (present or not). | at 6 month
  Binary (present or absent)
radiographic indications of radiolucency and pathologic root resorption (periapical or bifurcation) will be examined (present or not). | at 1 year
  Binary (present or absent)

CONTACTS AND LOCATIONS:
Overall Officials: ahmed m Elkhadem, Ass.Prof, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No